CLINICAL TRIAL: NCT05329298
Title: A Phase 1/2 Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of BPI-361175 in Subjects With Advanced Solid Tumors
Brief Title: A Phase 1/2 Study of BPI-361175 in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BTP-661411
Record Dates: First submitted 2022-03-31; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase I (Experimental): Patients will receive a single dose on Day 1, then after an 7-day wash-out period, repeated dosing, once daily will be initiated(Ia).
  Patients receive BPI-361175 PO. Cycles repeat every 28 days(Ib).
  Interventions: Drug: BPI-361175
- Phase II (Experimental): Patients receive BPI-361175 based on RP2D.
  Interventions: Drug: BPI-361175

INTERVENTIONS:
Drug: BPI-361175 — Subjects will receive BPI-361175 until disease progression

SUMMARY:
This is a phase I/II, open-label study to evaluate the safety, tolerability, pharmacokinetics and anti-tumor activity of BPI-361175 tablets in patients with advanced solid tumors including advanced Non-small cell Lung cancer (NSCLC).This is a three-stage study, consisting of Phase Ia dose escalation, Phase Ib dose expansion and pivotal Phase II Study. The pivotal Phase II study will be designed based on data generated from the Phase I studies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years old;
* Patients with histologically or cytologically confirmed diagnosis of inoperable locally advanced or recurrent/metastatic non-small cell lung cancer (NSCLC) with EGFR sensitive mutations. Patients must have progressed from or be intolerant to or be unfit for standard treatment, or the standard treatment does not exist;
* For dose expansion and Phase II, patients must be willing to provide tumor tissues (archived tumor tissue samples within 2 years or fresh tumor tissues) and/or blood samples for central lab testing;
* Measurable or evaluable disease;
* Adequate bone marrow, liver, and renal function.

Exclusion Criteria:

* Unstable, symptomatic primary CNS tumors/metastasis or leptomeningeal metastases which are not suitable for enrollment, as judged by investigators;
* Pregnancy or lactation;
* Other protocol specified criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase I: The adverse events (AEs) | Through the Phase I, approximately 24 months
  Safety and tolerability will be assessed by monitoring frequency, duration and severity of adverse events (AEs).
Phase I: Determine the recommended Phase II dose (RP2D) | Through the Phase I, approximately 24 months
  Number of subjects with dose limiting toxicity
Phase II: the objective response rate (ORR) | Through the Phase II, approximately 24 months
  The proportion of patients with complete response (CR) and partial response (PR) in all patients.

SECONDARY OUTCOMES:
Phase I: Evaluate the pharmacokinetics of BPI-361175 | Through the Phase I, approximately 24 months
  Blood plasma concentration
Phase I: the objective response rate (ORR) | Through the Phase I, approximately 24 months
  The proportion of patients with complete response (CR) and partial response (PR) in all patients.
Phase II: Disease control rate (DCR) | Through the Phase II, approximately 24 months
  The proportion of patients with CR, PR and stable disease (SD) in all patients.
Phase II: Progression free survival (PFS) | Through the Phase II, approximately 24 months
  The time from the first study dose to disease progression (PD) or death, whichever occurs first.
Phase II: Overall survival (OS) | Through the Phase II, approximately 24 months
  The time from the first study dose to death due to any cause.
Phase II: Duration of response (DOR) | Through the Phase II, approximately 24 months
  The time from the first CR or PR to the first PD or death due to any cause.
Phase II: The adverse events (AEs) | Through the Phase II, approximately 24 months
  Safety and tolerability will be assessed by monitoring frequency, duration and severity of adverse events (AEs).
Phase I: Disease control rate (DCR) | Through the Phase I, approximately 24 months
  The proportion of patients with CR, PR and stable disease (SD) in all patients.
Phase I: Progression free survival (PFS) | Through the Phase I, approximately 24 months
  The time from the first study dose to disease progression (PD) or death, whichever occurs first.
Phase I: Overall survival (OS) | Through the Phase I, approximately 24 months
  The time from the first study dose to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Ph.D, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China; Jianying Zhou, Ph.D, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (8):
- China (8):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan cancer hospital, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - the First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No